CLINICAL TRIAL: NCT00338533
Title: Endoscopic Goniotomy for Infantile Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Karen Joos, Associate Professor of Ophthalmology, Vanderbilt University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Vanderbilt IRB # 8542
Record Dates: First submitted 2006-06-15; First posted 2006-06-20 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Glaucoma
Keywords: childhood glaucoma
MeSH Terms: conditions — Glaucoma; Hydrophthalmos

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: endoscopic goniotomy — The goninotomy is performed through an endoscope; allowing the physician a better view of the structure within the eye

SUMMARY:
Glaucoma surgery is performed on children less than 3 years old for infantile glaucoma which untreated can cause blindness. Glaucoma is an uncontrolled high eye pressure in these children often due to incomplete development of the part of the eye which normally allows fluid to drain out of the eye. Two procedures are possible and equal in their success of lowering the eye pressure. However, one (the goniotomy procedure) is preferred since it takes 10 minutes rather than 1 hour (for the trabeculotomy procedure) to perform under general anesthesia. This is important in young children to reduce anesthesia exposure especially if both eyes need surgery. If the glaucoma has caused the cornea or front of the eye to become too cloudy, then the view is too poor to place a lens on the cornea and use a needle to perform the shorter procedure. However, a small endoscope which has been FDA approved for use in the eye will allow direct viewing of the area which needs treatment. A needle attached to this endoscope allows the shorter goniotomy to be performed rather than proceeding to the longer trabeculotomy procedure. The outcome measure of this study is anesthesia time and reduction in intraocular pressure .

DETAILED DESCRIPTION:
b. The standard examination under anesthesia initially will be performed including measuring the child's intraocular pressure, measuring dimensions of the eye, examining the front of the eye under the operating microscope, examining the portion of the eye where the fluid drains, evaluating the back of the eye with an ultrasound, and possible documentation with photographs.

When the diagnosis is confirmed by this examination, the eye or eyes will be carefully evaluated for their clarity. If a standard goniotomy procedure can not be done, then the endoscopic goniotomy will be performed. The procedure is identical with: cleaning the eyelid skin, using a speculum to open the eyelids, making a small cut into the cornea, and placing a viscoelastic substance into the eye to maintain its shape. The procedure then differs since the inserted needle is attached to the viewing endoscope. I will then view the inside of the eye on a TV monitor in addition to looking through the operating microscope. This will allow me to directly see the structures which I will need to cut. Normally, I depend upon looking through a lens placed on the cornea which must be fairly clear so that I can see to cut the structures in the standard procedure. The procedure should not take much longer than the standard goniotomy and the same amount of tissue will be cut as in a standard goniotomy. The needle is then removed. The remainder of the procedure is identical which includes placing a stitch in the corneal incision, adjusting the amount of fluid in the eye so the pressure is not too low or high, giving a dilating drop, giving a steroid and antibiotic injection around the eye, giving steroid ointment and an eye patch.

ELIGIBILITY:
Inclusion Criteria:

* childhood glaucoma with corneal edema unable to perform goniotomy

Exclusion Criteria:

* older than 3 years

Ages: 1 Week to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 1997-04; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure reduction | Postoperatively

SECONDARY OUTCOMES:
Clearing of corneal edema | Postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: karen Joos, MD, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- [Result] Joos KM, Shen JH. An ocular endoscope enables a goniotomy despite a cloudy cornea. Arch Ophthalmol. 2001 Jan;119(1):134-5. No abstract available. PMID 11146740